CLINICAL TRIAL: NCT00722345
Title: Can Exercise Consultation Increase Activity Levels and Improve Metabolic Markers in Obese Adolescents? A Pilot Study.
Brief Title: Exercise Consultation in Obese Youth
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: St. Justine's Hospital (Other)
Responsible Party: Dr. Celine Huot, Ste-Justine Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2162
Record Dates: First submitted 2008-07-23; First posted 2008-07-25 (Estimated); Last update posted 2008-07-25 (Estimated); Status verified 2005-06

CONDITIONS: Obesity
Keywords: Obesity; Physical activity; Adolescents; Exercise counseling intervention
MeSH Terms: conditions — Obesity; Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Placebo Comparator)
  Interventions: Behavioral: review of "Canada's Physical Activity Guide for Youth"
- 2 (Experimental)
  Interventions: Behavioral: Exercise consultation

INTERVENTIONS:
Behavioral: review of "Canada's Physical Activity Guide for Youth" — The contents of the exercise booklet was reviewed with each participant of the control group by the research fellow. Health Canada's "Canada's Physical Activity Guide for Youth" was used for the exercise booklet
  Arms: 1
Behavioral: Exercise consultation — The exercise consultation consisted of a one-to-one discussion designed to educate the participant, strengthen his/her motivation and develop realistic goals and strategies to promote physical activity based on the patient's stage of change. The consultation was based upon the standardized protocol previously published by Loughlan and Mutrie. The Consultation Guidelines describe the 5 steps involved in an exercise consultation, including: 1) discussing current & past activities; 2) reviewing the pros & cons of exercising; 3) discussing the barriers to exercising and strategies for overcoming them; 4) determining the social support available to the patient; and finally, 5) setting realistic, attainable short term and long term goals to enhance physical activity.
  Arms: 2

SUMMARY:
Exercise consultation, an intervention approach based on the transtheoretical model has been successful in promoting physical activity (PA) among adults. It is unknown whether this approach would be efficacious with youth. The purpose of this pilot study was to assess whether exercise consultation would increase PA levels and improve anthropometric measures and metabolic markers in obese adolescents.

ELIGIBILITY:
Inclusion Criteria:

* Adolescents
* BMI greater than or equal to the 95th percentile for age (2000 CDC growth charts)

Exclusion Criteria:

* Pregnancy
* Underlying medical condition, physical or cognitive disability that will impair individual's ability to participate in physical activity

Ages: 14 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 33 (Actual)
Dates: Start 2005-06; Primary Completion 2006-08 (Actual); Study Completion 2006-08 (Actual)

PRIMARY OUTCOMES:
Physical activity counts per minute (accelerometer data) | At baseline and at 3 months

SECONDARY OUTCOMES:
Stage of change | At baseline and at 3 months
Lipids | At baseline and at 3 months
Glucose | At baseline and at 3 months
Insulin | At baseline and at 3 months
Blood pressure | At baseline and at 3 months
Anthropometric mesures (height, weight, waist circumference, hip circumference) | At baseline and at 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Melanie Henderson, MD MSc FRCP, Principal Investigator — Ste-Justine Hospital/McGill University; Celine Huot, MD MSc, Principal Investigator — Ste-Justine Hospital/University of Montreal; Denis Daneman, MB BCh FRCP, Principal Investigator — University of Toronto; Janet Hux, MD SM, Principal Investigator — University of Toronto; Anthony Hanley, PhD, Principal Investigator — University of Toronto; Jennifer McGrath, PhD MPH, Principal Investigator — Concordia University, Montreal; Marie Lambert, MD, Principal Investigator — Ste-Justine Hospital/University of Montreal; Gillian L Booth, MD MSc, Principal Investigator — University of Toronto
Locations (1):
- Centre Hospitalier Universitaire Ste-Justine, Montreal, Quebec, Canada